CLINICAL TRIAL: NCT03051386
Title: Phase 2 Open-Label Safety and Immunogenicity Study of the Venezuelan Equine Encephalomyelitis (VEE) Vaccine, Live Attenuated, Dried, TC-83, NDBR 102, Lot 4, Run 3, as Primary Vaccination in Healthy Adult Subjects at Risk of Exposure to VEE Virus
Brief Title: Safety and Immunogenicity of Venezuelan Equine Encephalomyelitis Vaccine in Healthy Adults
Acronym: VEE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-13-04; IND 142 (Other: Food and Drug Administration); M-10510 (Other: IRB); FY15-12 (Other: USAMRIID)
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Venezuelan Equine Encephalomyelitis Virus Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VEE Vaccine (Experimental): 0.5 mL of VEE vaccine, Live, Attenuated TC-83, NDBR 102, Lot 4, Run 3
  Interventions: Biological: VEE Vaccine

INTERVENTIONS:
Biological: VEE Vaccine — 0.5 mL of VEE vaccine administered subcutaneously in the upper outer aspect of the triceps region.
  Other Names: TC-83

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of VEE vaccine, Live, Attenuated, dried TC-83, NDBR 102, Lot 4, Run 3, and collect data on the incidence of occupational VEE virus infection in vaccinated personnel.

DETAILED DESCRIPTION:
This protocol is replacing NCT00582504.

The study population will consist of USAMRIID and qualified extramural participants who are at risk of exposure to VEE virus. This study will be performed at the USAMRIID SIP Clinic. This open-label study represents a continuation of previous research conducted at USAMRIID. Subjects will be vaccinated with 0.5 mL of VEE vaccine, Live, Attenuated TC-83, NDBR 102, Lot 4, Run 3 subcutaneously in the upper outer aspect of the triceps region. Subjects will contacted the following day and weekly for 4 weeks to assess for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18-65 years old at time of consent.
2. Have VEE virus PRNT80 < 1:10.
3. If female of childbearing potential, must agree to have a serum pregnancy test on the same day before vaccine administration. (Exception: documented hysterectomy or ≥ 3 years of menopause.) The results must be negative. Females must agree not to become pregnant for 3 months after receipt of the vaccination.
4. Be considered at risk for exposure to VEE virus and who have submitted a Request for IND Vaccines for the VEE vaccine.
5. Sign and date the approved informed consent document and HIPAA Authorization.
6. Have in their charts:

   * medical history (including concomitant medications) within 60 days of planned first administration of vaccine
   * physical examination and laboratory tests within 1 year
   * previous chest radiograph results and electrocardiogram
7. Be medically cleared for participation by an investigator. Examinations or tests may be repeated at the discretion of the PI.
8. Be willing to return for all follow-up visits.
9. Agree to report any AEs that may or may not be associated with administration of the vaccine for at least 28 days after administration and agree to report all SAEs (for example, resulting in hospitalization) for the duration of the subject's participation in the study.
10. Agree to defer blood donation for 1 year after receipt of the vaccine.

Exclusion Criteria:

1. Have received VEE vaccine.
2. Have family history (first degree relative) of diabetes mellitus (any type), a personal or family history of gestational diabetes, a confirmed elevated fasting serum glucose test (> 125 mg/dL), or a hemoglobin A1c > 5.6%. (At the principal investigator's discretion, a subject may participate if the family history of diabetes is only of late onset in an elderly parent.)
3. Have clinically significant abnormal laboratory results (including evidence of hepatitis C, hepatitis B carrier state) or elevated liver function tests (two times the normal range or at the discretion of the PI).
4. Have a personal history of an immunodeficiency or received treatment with an immunosuppressive medication, such as systemically administered glucocorticoids (eg prednisone) within 1 month before planned administration of the vaccine or with other immunosuppressive therapies within 6 months of planned administration of the vaccine. Other immunosuppressive therapies include all cancer chemotherapeutic agents, drugs to prevent transplant rejection, interferons, monoclonal antibodies, protein kinase inhibitors, methotrexate, TNF (tumor necrosis factor) inhibitors, and any other drug determined to be immunosuppressive by the PI. Current administration of topical, inhalational, or intranasal glucocorticoids is not excluded.
5. Have confirmed HIV infection (antibody positivity).
6. Have a positive pregnancy test or a breastfeeding female.
7. Have any known allergies to components of the vaccine:

   * Neomycin sulfate
   * Guinea pig heart cells
   * Streptomycin
   * Human serum albumin
8. History of serious allergic reaction to guinea pigs or guinea pig products. (Subjects who have known allergies to guinea pigs will be evaluated. The vast majority of individuals who are allergic to guinea pigs are allergic to the dander from the animals. An individual with a past serious allergic reaction to guinea pigs will be excluded.)
9. Have administration of another vaccine or investigational product within 28 days of VEE vaccination.
10. Have any unresolved AE resulting from a previous immunization.
11. Have a medical condition that, in the judgment of the PI, would impact subject safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety: Occurrence of Serious Adverse Events and Adverse Events (SAEs and AEs) | 15 months
  Collect and assess safety data for VEE vaccine
Safety: Percentage of subjects with symptoms following VEE vaccination | 15 months
  Collect and assess safety data for VEE vaccine
Safety: Percentage of subjects with each AE, system organ class of AE, severity, and association with vaccination | 15 months
  Collect and assess safety data for VEE vaccine

SECONDARY OUTCOMES:
Immunogenicity: Percentage of subjects who develop titers of >1:20 | 15 months
  Percentage of subjects who develop titers of ≥ 1:20 as determined by PRNT80 after VEE vaccination at each scheduled time point for which blood samples are taken and over the entire study period to study completion.
Immunogenicity: Geometric Mean PRNT80 Titers of subjects | 15 months
  Geometric mean PRNT80 titers of subjects at each scheduled time point for which blood samples are taken and over the entire study period to study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B. Reisler, MD, MPH, Principal Investigator — USAMRIID
Locations (1):
- Special Immunizations Program, Division of Medicine, USAMRIID, Fort Deterick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No